CLINICAL TRIAL: NCT00564525
Title: Evaluation of the Efficacy of Amitriptyline in Children With Abdominal Pain of Non-Organic Origin
Brief Title: Study of Medication for Functional Abdominal Pain in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: American College of Gastroenterology (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-12430
Record Dates: First submitted 2007-11-27; First posted 2007-11-28 (Estimated); Last update posted 2007-11-28 (Estimated); Status verified 2007-11

CONDITIONS: Functional Gastrointestinal Disorders
Keywords: children; abdominal pain; amitriptyline
MeSH Terms: conditions — Gastrointestinal Diseases; Abdominal Pain | interventions — Amitriptyline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental): Amitriptyline given
  Interventions: Drug: Amitriptyline

INTERVENTIONS:
Drug: Amitriptyline — Medication taken for 4 weeks
  Other Names: Other names include: Elavil, Trepiline and Laroxyl.
  Arms: 2
Drug: Placebo — Medication taken for 4 weeks
  Arms: 1

SUMMARY:
The purpose of this study is to determine where amitriptyline is effective in the treatment of functional abdominal pain in children.

DETAILED DESCRIPTION:
Recurrent gastro-intestinal complaints constitute one of the most common reasons for medical consultation among daycare and school children. Studies suggest an association between childhood functional abdominal pain and psychiatric disorders. Although most children with mild symptoms are mostly managed by reassurance and simple measures, a large range of interventions such as dietary changes, use of antidepressant and medications are being widely used with little evidence to suggest their effectiveness. In view of the high prevalence of this disorder and the lack of pediatric scientific evidence on extensively used drug therapies there is critical need to develop trials of all suggested pharmacologic interventions in children with functional pain disorders. This study has the potential to fill a critical void in pediatric gastroenterology.

The main objective of this study is to evaluate the impact of the medication (amitriptyline) on symptoms of patients with abdominal pain of non-organic origin.

Our hypotheses are that amitriptyline results in adequate relief of symptoms in children with functional abdominal pain and that is more effective than placebo in controlling pain.

This is a randomized, double masked placebo controlled study, using standard current measures and diagnostic criteria to address the question whether the treatment with amitriptyline is efficacious, and that leads to an improvement in severity of the symptoms for which the patient sought medical attention.

The study is conducted on a group of children (eight to eighteen years) suffering from functional abdominal pain. The study population is randomly assigned (by chance) into 2 groups (half of the patients receive drug and half of patients receive a non-acting drug-placebo). Each individual will randomly receive the medication or placebo at night time for 4 weeks. In order to qualify for the study the patients have to complete one week on baseline questionnaires to assess their symptoms and have to be diagnosed with a condition associated with functional abdominal pain by the investigators. The patient will complete initial questionnaires and end of the study questionnaires as well as daily questionnaires to assess the symptoms. At the end of the study both groups will be compared to establish differences.

ELIGIBILITY:
Inclusion Criteria:

* Age 8 to 17 years
* Diagnosis of functional abdominal pain or irritable bowel syndrome made by a pediatric gastroenterologist according to Rome II criteria
* Mean daily intensity of pain of 25 mm in the week prior to the initiation of the study, based on the Word-Graphic Rating Scale continuous score
* Following evaluation in the six months prior to the study: normal EKG and laboratory tests including complete blood count, erythrocyte sedimentation rate, albumin, serum amylase, lipase, liver enzymes, urine analysis, stool examination for occult blood and ova and parasites. Urinary culture will be obtained if the symptoms or urinalysis suggest the possibility of a urinary infection,
* Normal lactose breath test or history of lack of resolution of symptoms on a lactose-free diet
* Consenting parents
* Patient assent

Exclusion Criteria:

* Inclusion criteria not met
* Evidence of organic gastrointestinal disease, hepatic disorders, urinary or cardiac disease, seizures, blood dyscrasias, glaucoma
* History of allergic reaction to amitriptyline
* Patients receiving barbiturates, cimetidine, neuroleptics, monoamine oxidase inhibitors, sympathomimetic agents or quinidine
* Children below the 5th percentile for weight or height
* Hemoccult positive stools

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2002-10; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Patient report on wether amitriptyline therapy resulted in adequate relief of symptoms | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Saps, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Children's Memorial Hospital, Chicago, Illinois, United States